CLINICAL TRIAL: NCT07067918
Title: Effects of Upper and Lower Body Plyometric Training on Kickboxing Anaerobic Speed Test Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Abdullah Demirli, Assistant Professor, Ph.D., Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ETU-BAEK-2025-02-10
Record Dates: First submitted 2025-07-07; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Effects of Upper and Lower Body Plyometric Training on Anaerobic Performance in Combat Sport Athletes; Sport-specific Anaerobic Performance in Elite Male Kickboxers
Keywords: Plyometrics; anaerobic performance; sport-specific; KAST; combat sports

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to one of two parallel groups: upper-body plyometric training or lower-body plyometric training. Both groups continued their standard kickboxing training while following a 12-week intervention protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 - Upper Body Plyometric Group (Experimental): Participants in this group completed a 12-week upper-body plyometric training program including medicine ball throws, plyometric push-ups, and explosive arm drills.
  Interventions: Other: Upper Body Plyometric Training
- Arm 2 - Lower Body Plyometric Group (Experimental): Participants in this group followed a 12-week lower-body plyometric training protocol including squat jumps, depth jumps, and lateral hurdle jumps.
  Interventions: Other: Lower Body Plyometric Training

INTERVENTIONS:
Other: Upper Body Plyometric Training — Upper Body Plyometric Training - Intervention Description:
  A 12-week upper-body plyometric training protocol designed to enhance explosive upper-extremity power in elite male kickboxers. Exercises included medicine ball chest passes, overhead throws, plyometric push-ups, clap push-ups, and rotational medicine ball throws. Training was performed three times per week (20-30 minutes per session) in addition to regular kickboxing practice.
  Arms: Arm 1 - Upper Body Plyometric Group
Other: Lower Body Plyometric Training — Lower Body Plyometric Training - Intervention Description:
  A 12-week lower-body plyometric training program targeting explosive leg strength and anaerobic performance in elite male kickboxers. The program included countermovement jumps, squat jumps, lateral hurdle jumps, plyometric bounding, tuck jumps, and depth jumps. Sessions were conducted three times per week (20-30 minutes each), alongside regular kickboxing training.
  Arms: Arm 2 - Lower Body Plyometric Group

SUMMARY:
This study examined the effects of two different types of jump training-one focused on the upper body and the other on the lower body-on the athletic performance of elite male kickboxers. Over a 12-week period, athletes followed specific exercise programs designed to increase explosive power in either the arms or the legs, while continuing their normal kickboxing training.

Researchers used a special performance test called the Kickboxing Anaerobic Speed Test (KAST), which measures how fast and powerfully athletes can punch and kick over a short time. The results showed that while both training methods improved performance, the group that did lower-body jump training (e.g., leg-focused exercises) showed greater gains. This suggests that strong and explosive legs play a key role in powerful strikes and quick movements in kickboxing.

In summary, lower-body jump training is more effective than upper-body jump training in improving sport-specific speed and power in elite male kickboxers.

DETAILED DESCRIPTION:
This study aimed to compare the effects of upper- and lower-body plyometric training on anaerobic performance in elite male kickboxers. Thirty-two national-level athletes were randomly assigned to one of two training groups: one focusing on upper-body exercises (e.g., medicine ball throws, explosive push-ups), and the other on lower-body exercises (e.g., squat jumps, depth jumps). Both groups continued their regular kickboxing training while performing the additional plyometric training three times per week over 12 weeks.

Anaerobic performance was measured using the Kickboxing Anaerobic Speed Test (KAST), which assesses sport-specific punching and kicking combinations under time pressure. Pre- and post-intervention assessments included KAST best time, total time, and fatigue index.

The results showed that while both training programs improved performance, the lower-body training group achieved greater improvements in speed and power. These findings suggest that explosive strength in the legs plays a critical role in kickboxing performance, especially for actions like kicking and stabilizing during punching.

This trial highlights the importance of lower-body plyometric exercises for enhancing combat sport performance and may help coaches design more effective training plans for elite-level kickboxers.

ELIGIBILITY:
Inclusion Criteria:

* Male participants aged 18 to 35 years
* At least 5 years of structured kickboxing training
* Active competition status within the last 3 years
* Minimum of one national or international medal in the past 2 years
* Provided written informed consent

Exclusion Criteria:

* No formal kickboxing training history
* No competitive activity in the last 3 years
* No documented medal success at national or international level
* Failure to meet informed consent or ethical participation requirements

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2025-02-15 (Actual); Primary Completion 2025-05-22 (Actual); Study Completion 2025-06-10 (Actual)

PRIMARY OUTCOMES:
Best score time in the Kickboxing Anaerobic Speed Test (KASTbest) | Measured at baseline and 12 weeks
  The best completion time for a five-technique striking sequence performed at maximum intensity. A lower score indicates better anaerobic performance.
Performance Decrement Index (PDI) | Measured at baseline and 12 weeks
  The ratio between the athlete's best performance time and cumulative performance across sets, used to assess fatigue resistance during high-intensity intermittent effort.

SECONDARY OUTCOMES:
Total time in the Kickboxing Anaerobic Speed Test (KASTtotal) | Measured at baseline and 12 weeks
  The total time required to complete five sets of the KAST striking protocol. A lower time indicates better anaerobic endurance.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University Cerrahpaşa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No